CLINICAL TRIAL: NCT02583490
Title: Low Pulse Amplitude Focal Electroconvulsive Therapy
Brief Title: Low Pulse Amplitude Focal ECT (LAP Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Nagy Adel Youssef, Associate Professor, Psychiatry and Health Behavior, Augusta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Low Pulse Amplitude Focal ECT
Record Dates: First submitted 2015-10-13; First posted 2015-10-22 (Estimated); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Depression
Keywords: Electroconvulsive Therapy; Low Pulse Amplitude Focal Electroconvulsive Therapy; ECT; Depression; Suicidal Ideation
MeSH Terms: conditions — Depression; Suicidal Ideation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low Pulse Amplitude ECT (LAP) (Experimental): Right Unilateral LAP ECT
  Interventions: Device: spectrum 5000Q ECT device (RUL LAP ECT)
- standard Right Unilateral ECT (Active Comparator): standard Right Unilateral ECT
  Interventions: Device: spectrum 5000Q ECT device (RUL ECT)

INTERVENTIONS:
Device: spectrum 5000Q ECT device (RUL ECT)
  Arms: standard Right Unilateral ECT
Device: spectrum 5000Q ECT device (RUL LAP ECT)
  Arms: Low Pulse Amplitude ECT (LAP)

SUMMARY:
This protocol proposes a pilot randomized clinical trial to examine whether Low Pulse Amplitude Focal ECT (LAP) has a more favorable cognitive profile compared to conventional unilateral ECT and that it has similar effects as traditional ECT in reducing suicidality. The study will enroll 10 patients recruited from the Medical College of Georgia (at Georgia Regents University/Augusta University, GRU/AU) as the only site of the study. Eligible participants will be randomly assigned (1:1 ratio) to receive a course of either RUL LAP ECT, or conventional RUL ECT.

DETAILED DESCRIPTION:
Lower amplitude ECT (LAP) has been shown to induce seizures of adequate duration in a single titration session. This current study is hypothesized to increase stimulation focality, thus hypothetically minimizing cognitive side effects.

The central hypothesis is that LAP has significantly less cognitive adverse effects compared to conventional Right Unilateral (RUL) ECT.

The study will enroll 10 patients recruited from Medical College of Georgia. Patients referred to ECT service in the Medical College of Georgia usually occurs from clinical services and private physicians and the study will recruit patients who are clinically indicated to do ECT. Eligible participants will be randomly assigned (1:1 ratio) to receive a course of either RUL LAP ECT, or conventional RUL ECT.

ELIGIBILITY:
Inclusion Criteria:

* Patients in whom ECT therapy is clinically indicated
* Males or females patients over 20 years of age
* Current DSM-IV criteria for major depressive episode
* Montgomery-Asberg depression rating scale (MADRS) greater than or equal to 20
* Use of effective method of birth control for women of child-bearing capacity
* Patient is medically stable
* No anticipated need to alter psychotropic medications for the duration of the study
* Ability of patient to fully participate in the informed consent process

Exclusion Criteria:

* Unstable or serious medical condition that substantially increases risks of ECT or of cognitive impairment
* Substance use disorders within 1 week of randomization
* History of neurological disorder, epilepsy, stroke, brain surgery, metal in the head, history of known structural brain lesion that is deemed to affect cognition or safe ECT treatment
* Vagal Nerve Stimulator implanted
* Female patients who are pregnant or plan to be pregnant during the study breast-feeding
* Implanted devices that make ECT unsafe, or a skull defect
* Significant cognitive impairment (Mini-Mental State Examination (MMSE) less than 24)
* ECT in the past 1 months
* Benzodiazepine use will be limited to no more than 3 mg per day of lorazepam or its equivalents. Antidepressants and antipsychotics will be held constant during the ECT course of the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Memory (cognitive side effects) | From Baseline to end of acute course (typically after 4 weeks)
  Measured by Autobiographic Memory Interview-Short form (AMI-SF, primary outcome)
Time to reorientation | From Baseline to end of acute course (typically after 4 weeks)
  Measured by Time to Orientation Test (TRO, primary outcome)

SECONDARY OUTCOMES:
Resilience | From Baseline to end of acute course (typically after 4 weeks)
  Connor-Davidson Resilience Scale
Suicidal Ideation | From Baseline to end of acute course (typically after 4 weeks)
Depression | From Baseline to end of acute course (typically after 4 weeks)
  used to determine remission status; measured by Montgomery-Åsberg Depression Rating Scale (MADRS)
Depression | From Baseline to end of acute course (typically after 4 weeks)
  Patient Health Questionnaire (PHQ 9)
Trauma symptoms | From Baseline to end of acute course (typically after 4 weeks)
  PTSD Checklist

CONTACTS AND LOCATIONS:
Overall Officials: Nagy Youssef, MD, Principal Investigator — Augusta University
Locations (1):
- Medical Colleage of Georgia, Augusta University, Evans, Georgia, United States

REFERENCES:
- [Result] Youssef NA, Ravilla D, Patel C, Yassa M, Sadek R, Zhang LF, McCloud L, McCall WV, Rosenquist PB. Magnitude of Reduction and Speed of Remission of Suicidality for Low Amplitude Seizure Therapy (LAP-ST) Compared to Standard Right Unilateral Electroconvulsive Therapy: A Pilot Double-Blinded Randomized Clinical Trial. Brain Sci. 2019 Apr 29;9(5):99. doi: 10.3390/brainsci9050099. PMID 31035665
- [Derived] Youssef NA, Dhanani S, Rosenquist PB, McCloud L, McCall WV. Treating Posttraumatic Stress Disorder Symptoms With Low Amplitude Seizure Therapy (LAP-ST) Compared With Standard Right Unilateral Electroconvulsive Therapy: A Pilot Double-Blinded Randomized Clinical Trial. J ECT. 2020 Dec;36(4):291-295. doi: 10.1097/YCT.0000000000000701. PMID 33215889